CLINICAL TRIAL: NCT07352891
Title: Digital Remote Management for Care and Continuous Optimization Versus Usual Care to Improve Prognosis in Patients With Heart Failure With Reduced Ejection Fraction (DigiCare-HFrEF): A Multicentre, Randomised, Controlled Trial
Brief Title: Digital Remote Management for Care and Continuous Optimization Versus Usual Care to Improve Prognosis in Patients With Heart Failure With Reduced Ejection Fraction
Acronym: DigiCare-HFrEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang sheng Ma (Other)
Responsible Party: Sponsor-Investigator, Chang sheng Ma, Director of cardiology department, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS2025289
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual Care with guideline-recommended outpatient follow-up. No platform-based risk stratification or decision support is provided.
- Digital Remote Management (Experimental): Participants will use a digital remote-management platform to report symptoms and key physiologic variables (e.g., blood pressure and body weight). The platform applies a predefined risk-stratification algorithm and provides clinician-facing decision support for GDMT titration and congestion management. A comprehensive management for core health metrics will also be provided. Clinicians review and confirm recommendations before they are communicated to patients.
  Interventions: Other: Digital Remote Management

INTERVENTIONS:
Other: Digital Remote Management — Participants will use a digital remote-management platform to report symptoms and key physiologic variables (e.g., blood pressure and body weight). The platform applies a predefined risk-stratification algorithm and provides clinician-facing decision support for GDMT titration and congestion management. A comprehensive management for core health metrics will also be provided. Clinicians review and confirm recommendations before they are communicated to patients.
  Arms: Digital Remote Management

SUMMARY:
DigiCare-HFrEF is an investigator-initiated, multicentre, randomised, open-label, endpoint-blinded, superiority trial designed to evaluate whether a structured digital remote-management platform can improve clinical outcomes in patients with heart failure with reduced ejection fraction (HFrEF) after hospital discharge. Eligible adults with LVEF ≤40% within past 3 months, NYHA class II-IV, and elevated natriuretic peptides (NT-proBNP >2500 pg/mL or BNP >600 pg/mL) will be randomly assigned (1:1) to digital remote management or to usual care. In the intervention arm, patients will report symptoms and key physiologic measures (e.g., blood pressure and body weight) via the platform; an algorithm will perform risk stratification and generate guideline-directed medical therapy (GDMT) optimisation suggestions and decongestion prompts, as well as a comprehensive management for core health metrics, which are reviewed and confirmed by clinicians before implementation. The primary endpoint is the composite of cardiovascular death or first heart-failure event (hospitalisation or urgent visit for heart failure) at 12 months.

DETAILED DESCRIPTION:
"Heart failure with reduced ejection fraction (HFrEF) remains associated with high rates of early post-discharge events. In routine practice, timely optimisation of guideline-directed medical therapy (GDMT) and early recognition of haemodynamic deterioration are frequently limited by infrequent follow-up, delayed access to physiologic data, and variability in patient self-management.

DigiCare-HFrEF will enroll hospitalised patients with confirmed HFrEF and randomise them to either:

1. digital remote management based on an integrated platform that supports daily symptom and vital-sign reporting, algorithm-driven risk stratification, and clinician-reviewed decision support for GDMT titration and congestion management, plus standard guideline-based care; or
2. usual care with medical therapy and regular follow-up.

Randomisation will be performed through a central web-based system with stratification by participating centre and age (≤65 vs >65 years). Given the nature of the intervention, treatment allocation is open label; however, outcome assessment and event adjudication will be performed by independent personnel blinded to treatment assignment. Participants will be followed with standardised remote assessments at 1 and 6 months and face-to-face visits at 3 and 12 months. The trial will test whether a closed-loop digital care pathway-continuous monitoring, rapid risk-informed evaluation, and standardised responses with clinician oversight-reduces major clinical events and improves GDMT optimisation."

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years.
2. Hospitalised at a secondary or tertiary hospital with established heart failure care capacity.
3. Diagnosed with HFrEF within the past 3 months according to the 2022 ACC/AHA/HFSA guideline diagnostic pathway, including: LVEF ≤40% by echocardiography; typical heart-failure symptoms and/or signs; and exclusion of non-HF causes of symptoms.
4. NT-proBNP >2500 pg/mL or BNP >600 pg/mL.
5. NYHA functional class II-IV.
6. Written informed consent provided."

Exclusion Criteria:

1. Absolute contraindication to heart failure pharmacotherapy.
2. History of heart transplantation or currently on a transplant waiting list.
3. Receiving or planning implantation of a left ventricular assist device.
4. Pregnant or breastfeeding women.
5. Organ transplantation within the past 12 months.
6. Unable to use the remote management platform as required (e.g., cognitive impairment or lack of caregiver support).
7. Unable to perform blood pressure or body-weight monitoring (e.g., severe limb disability).
8. Unable to express willingness or comply with follow-up requirements (e.g., unable to use internet-enabled devices).
9. Estimated life expectancy <1 year.
10. Any other condition judged by the investigator to make the patient unsuitable for participation."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death or first heart failure event | 12 months after randomization
  hospitalisation or urgent visit for heart failure

SECONDARY OUTCOMES:
Change in hear failure GDMT score (ΔGDMT) from baseline to 3 months | 3 months after randomization
  The Guideline-Directed Medical Therapy (GDMT) Score is a modified heart-failure pharmacotherapy score based on five medication classes:
  1. angiotensin-converting enzyme inhibitors or angiotensin receptor blockers (ACEi/ARB),
  2. angiotensin receptor-neprilysin inhibitor (ARNI),
  3. beta-blockers (BB),
  4. mineralocorticoid receptor antagonists (MRA), and
  5. sodium-glucose cotransporter-2 inhibitors (SGLT2i).
  Dosing levels are scored as follows:
  * ACEi/ARB: 0 = none; 0 = <50% target dose; 1 = ≥50% target dose.
  * ARNI: 0 = none; 1 = <50% target dose; 2 = ≥50% target dose.
  * Beta-blocker: 0 = none; 1 = <50% target dose; 2 = ≥50% target dose.
  * MRA: 0 = none; 1 = <50% target dose; 2 = ≥50% target dose.
  * SGLT2 inhibitor: 0 = none; 2 = therapeutic dose (no low-dose category). The total GDMT Score ranges from 0 to 9, with higher scores indicating more complete, optimized, and guideline-concordant HF medical therapy.
First heart failure hospitalization | 3 months after randomization
First urgent visit for heart failure | 3 months after randomization
Total heart failure hospitalizations | 3 months after randomization
Total urgent visits for heart failure | 3 months after randomization
First cardiovascular hospitalization | 3 months after randomization
First all-cause hospitalization | 3 months after randomization
All-cause mortality | 3 months after randomization
First heart failure hospitalization | 12 months after randomization
First urgent visit for heart failure | 12 months after randomization
Total heart failure hospitalizations | 12 months after randomization
Total urgent visits for heart failure | 12 months after randomization
First cardiovascular hospitalization | 12 months after randomization
First all-cause hospitalization | 12 months after randomization
All-cause mortality | 12 months after randomization
Change in NT-proBNP from baseline | 12 months after randomization
Change in functional capacity (6-minute walk distance) | 12 months after randomization
Change in KCCQ score | 12 months after randomization
  The Kansas City Cardiomyopathy Questionnaire-23 (KCCQ-23) is a 23-item patient-reported outcome measure of heart-failure-specific health status (symptoms, physical and social limitations, and quality of life). Each item is rated on a 5-point Likert scale (1 = extremely limited to 5 = not at all limited; response options such as "limited for other reasons or did not do this activity" are treated as missing). Domain scores are transformed to a 0-100 scale, and the overall summary score ranges from 0 to 100, with higher scores indicating better health status and fewer symptoms.
Change in MLHFQ score | 12 months after randomization
  The Minnesota Living With Heart Failure Questionnaire (MLHFQ) is a 21-item instrument assessing heart-failure-related quality of life. Each item is scored from 0 ("no impact") to 5 ("very much"). The total score ranges from 0 to 105, with higher scores indicating worse quality of life.
Change in EQ-5D-5L score | 12 months after randomization
  The EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) describes health status in five domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each rated on 5 levels (1 = no problems to 5 = extreme problems). A utility index score is derived using the Chinese value set, with values ranging approximately from -0.281 to 1.000, and an accompanying visual analogue scale (VAS) score ranging from 0 to 100, where higher scores on both the index and the VAS indicate better health status.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, China, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing, China, Beijing
  - The First Affiliated Hospital of Dalian Medical University, Dalian, China, Dalian
  - The First Hospital of Jilin University, Changchun, China, Jilin
  - The Second Affiliated Hospital of Nanchang University, Nanchang, China, Nanchang
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China, Shanghai

IPD SHARING:
Plan to Share IPD: No